CLINICAL TRIAL: NCT05122897
Title: Temporary push-on Rings of Antimicrobial Alloys for Transmucosal Implant Abutment Systems: a Randomized Clinical Study on Early and Mature Biofilm Formation
Brief Title: Investigation of Biofilm Formation on Temporary push-on Rings of Implant Crowns
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: ITI International Team for Implantology, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 2021-D0061; ex21Zitzmann
Record Dates: First submitted 2021-11-03; First posted 2021-11-17 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Dental Plaque; Oral Biofilm; Peri-implantitis
Keywords: Titanium-6Aluminum-7Niobium alloy; Pagalinor; transmucosal implant abutment; implant crowns; temporary push-on rings; Variobase abutments
MeSH Terms: conditions — Dental Plaque; Peri-Implantitis

STUDY DESIGN:
Intervention Model Description: All patients enrolled in the current investigation will wear both the test and control ring material for a within-subject comparison. Ideally, biofilm sampling can be performed in a split mouth design (randomly allocated materials within subjects) with one patient having two implants for placing the test and the control material at the same time. In addition, patients providing one implant, will receive test and control push-on rings in a randomly assigned order, so that both materials are assessed in a consecutive manner.
Who Masked: Participant, Investigator
Masking Description: Double-blinded with the patient not knowing which material is placed, and the investigator and laboratory technicians have no information about the ring material.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pagalinor®2 (PA) test arm (Experimental): All patients will wear both the test and control ring material for a within-subject comparison. Ideally, biofilm sampling can be performed in a split mouth design (randomly allocated materials within subjects) with one patient having two implants for placing the test and the control material at the same time. In addition, patients providing one implant, will receive test and control push-on rings in a randomly assigned order, so that both materials are assessed in a consecutive manner.
  Interventions: Device: Rings made of PA (test)
- Titanium-6Aluminum- 7Niobium alloy (TAN) control arm (Active Comparator): All patients will wear both the test and control ring material for a within-subject comparison. Ideally, biofilm sampling can be performed in a split mouth design (randomly allocated materials within subjects) with one patient having two implants for placing the test and the control material at the same time. In addition, patients providing one implant, will receive test and control push-on rings in a randomly assigned order, so that both materials are assessed in a consecutive manner.
  Interventions: Device: Rings made of TAN (control)

INTERVENTIONS:
Device: Rings made of PA (test) — Rings made of PA (test) 0.2mm in thickness are pushed on the conical titanium base (abutment) of implant crowns and are removed and replaced after 48h, 2 weeks and 3 months for quantification of the bacterial biofilm. Test rings are applied in a split-mouth design provided that 2 implants are present (total of 4 months study period), or one after the other when only 1 implant is present (total of 8 months study period).
  Arms: Pagalinor®2 (PA) test arm
Device: Rings made of TAN (control) — Rings made of TAN (control) 0.2mm in thickness are pushed on the conical titanium base (abutment) of implant crowns and are removed and replaced after 48h, 2 weeks and 3 months for quantification of the bacterial biofilm. Control rings are applied in a split-mouth design provided that 2 implants are present (total of 4 months study period), or one after the other when only 1 implant is present (total of 8 months study period).
  Arms: Titanium-6Aluminum- 7Niobium alloy (TAN) control arm

SUMMARY:
This in-vivo study investigates early (48h), mature (2 weeks) and long-term (3 months) biofilm formation and composition on temporary push-on cones (exchangeable conical rings) made of noble-alloy-based materials (Pagalinor, PA) in comparison to Titanium-6Aluminum-7Niobium alloy (TAN) presently used in the transmucosal portion of dental implant abutments.

DETAILED DESCRIPTION:
Oral biofilm (dental plaque) consists of bacteria and their metabolic products as well as saliva components and food residues. It is recognizable as a tough and structured coating on teeth and artificial surfaces within the oral cavity. Plaque development is a physiological process that begins immediately after cleaning of the oral surface. If the biofilm is not removed by daily oral hygiene, it continues to mature while changing the structure and its microbial composition.

Implant restorations comprise the osseous implant portion predominantly manufactured from titanium alloys, the transmucosal implant portion (in most implant systems as a separate abutment), and the clinical crown, which is in most systems extraorally cemented on an abutment and screw-retained onto the implant. According to current knowledge, microbial colonization of the implant abutment surface plays a significant role in the aetiology of peri-implantitis.

This study investigates the antibacterial potential of a temporary push-on cone (conical ring) that could reduce the risk of bacterial related peri-implant diseases due to decreased biofilm susceptibility, compared to current available transmucosal materials, in the short- and long-run. The test material Pagalinor®2 (PA) is an established material in dental medicine and has proven to accumulate least biofilm in an in-vivo biofilm sampling model using removable splints. The control material consists of the current transmucosal implant abutment material Titanium-6Aluminum- 7Niobium alloy (TAN). The push-on rings are designed for repeated application along the transmucosal implant abutment portion with high precision fit and will allow biofilm sampling in the natural implant environment. Profound insight into the native homeostasis of biofilm formation will be obtained and therefore enhance the knowledge about long-term tissue response.

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent signed by the subject
* Presence of one or more bone level titanium implant prior to insertion of the final restoration
* No systemic illness
* No heavy smoking (smoking <10 cigarettes/day)
* No pregnancy
* No active periodontitis (probing pocket depth ≤4 mm)
* No pharmacological treatment or antibiotic therapy during or up to three months before the study

Exclusion Criteria:

* Systemic illness (e.g. Diabetes)
* Heavy smoking (smoking >10 cigarettes/day)
* Known or suspected non-compliance, drug or alcohol abuse
* Pregnancy
* Active periodontitis (probing pocket depth >4 mm)
* Pharmacological treatment or antibiotic therapy during or up to three months before the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2022-01-11 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Change in total bacterial load formed on the removable rings of each material | at 48 hours after ring placement, 2 weeks after ring placement and 3 months after ring placement
  Quantification of the bacterial load formed on the removable rings of each material by quantitative real-time PCR (qPCR) using primers specific to highly conserved regions of bacterial 16S rRNA genes.

SECONDARY OUTCOMES:
Change in bacterial composition (taxonomic diversity) between different materials at various time points by using metagenomic sequencing analysis | at baseline, 2 weeks after ring placement and 10 weeks after ring placement
  To assess differences in bacterial composition (taxonomic diversity) between different materials at various time points by Illumina MiSeq sequencing. The taxonomy of each 16S rRNA gene sequence will be analyzed by Ribosomal Database Project (RDP) Classifier (http://rdp.cme.msu.edu/) against the SILVA (SSU123) 16S rRNA database using a confidence threshold of 70%.
Change in probing pocket depth (PPD) in mm | at baseline, 2 weeks after ring placement and 10 weeks after ring placement
  Change in probing pocket depth (PPD) to investigate the inflammatory tissue response
Change in bleeding on probing (BoP) | at baseline, 2 weeks after ring placement and 10 weeks after ring placement
  Recording bleeding on probing (BoP) to investigate the inflammatory tissue response
Change in noninvasive laser doppler flowmetry | at baseline, 2 weeks after ring placement and 10 weeks after ring placement
  Change in noninvasive laser doppler flowmetry to to measure the blood flow of mucosa next to the ring
Change in the cells of the peri-implant soft tissue | at 2 weeks after ring placement
  To investigate the attachment of peri-implant soft tissues to implant materials, fibroblasts and junctional epithelial cells markers will be analysed using real-time quantitative PCR (RT-qPCR).

CONTACTS AND LOCATIONS:
Overall Officials: Nicola U. Zitzmann, Prof. Dr., Principal Investigator — University Center for Dental Medicine Basel
Locations (1):
- UZB (University Center for Dental Medicine Basel), Basel, Switzerland